CLINICAL TRIAL: NCT02604914
Title: 1) To Identify the Concentration of CD That Provides Optimal Bioavailability of a Concomitant Fixed Concentration of LD Infused SC Continuously; 2) To Compare the Bioavailability of the Optimal LD/CD Solution to That of LD/CD Intestinal Gel
Brief Title: A Sequential Two-Part, Open-Label Study in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ND0612-005
Record Dates: First submitted 2015-11-03; First posted 2015-11-16 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ND0612L (LD/CD solution) (Experimental): 3 doses of the investigational ND0612L (LD/CD solution) for subcutaneous (SC) infusion 0.24ml per hour.
  Interventions: Drug: ND0612
- ND0612H (LD/CD solution) (Experimental): 3 doses of the investigational ND0612H (LD/CD solution) for subcutaneous (SC) infusion 0.64ml per hour.
  Interventions: Drug: ND0612
- LCIG (Levodopa-carbidopa intestinal gel) (Active Comparator): Active Comparator: LCIG subjects who completed the ND0612H arm will be administered with 3 doses of LCIG, directly to the jejunum.
  Interventions: Drug: LCIG

INTERVENTIONS:
Drug: ND0612 — Subcutaneous solution
  Other Names: (Levodopa-Carbidopa solution)
  Arms: ND0612H (LD/CD solution); ND0612L (LD/CD solution)
Drug: LCIG — Intrajejunal Gel
  Other Names: (Levodopa-Carbidopa Intestinal Gel)
  Arms: LCIG (Levodopa-carbidopa intestinal gel)

SUMMARY:
An Open-Label Study in Healthy Male and Female Subjects to Identify the Concentration that Provides Optimal Bioavailability of Levodopa Infused Subcutaneously via a Pump System; and to Compare the Bioavailability of Levodopa/Carbidopa Solution to that of Levodopa/Carbidopa Intestinal Gel (LCIG), Infused via a Naso-Jejunal Tube

DETAILED DESCRIPTION:
Part 1: This is a single centre, open-label design with 2 study arms (ND0612H and ND0612L), in 24 subjects that will receive the ND0612L or ND0612H regimens. Part of the subjects will also participate in Part 2 of the study. Within each study arm, subjects will receive 3 doses of the investigational LD/CD solution for subcutaneous (SC) infusion. Study drug will be administered for 24 -30 hours as a subcutaneous (SC) infusion to the lower abdomen. Then subjects will be readmitted for Part 2. Part 2: This is a single centre, open-label design with 3 treatment arms to which 15 subjects who completed the ND0612H arm of Part 1 ND0612-005a will be allocated in a randomised manner. Within each treatment arm subjects will receive 2 out of 3 doses of LCIG infused for 16 hours directly to the jejunum. Subjects will be discharged from the clinic 24 hours after the end of the last infusion

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Part 1 ND0612-005a:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age 40 to 65 years of age
3. Body mass index of 18.0 to 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study (Part 1 only for subjects assigned to ND0612L and Part 1 and Part 2 for subjects assigned to ND0612H)
5. Must provide written informed consent
6. Area of administration to be evaluable for local skin reaction (normal skin without skin burns, scars or large tattoos in the area of administration)
7. Must agree to use an adequate method of contraception

Inclusion Criteria: Part 2 ND0612-005b:

1. Subjects who were dosed with ND0612H (any replacements subjects enrolled in Part 2 will be dosed with the optimal LD/CD concentration of ND0612H after completion of Part 2).

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
7. Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at admission)
8. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1)
9. Positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
10. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
12. History of cardiovascular, renal, hepatic, chronic respiratory or GI disease as judged by the investigator
13. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
14. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
15. Donation or loss of greater than 400 mL of blood within the previous 3 months
16. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol, hormone replacement therapy and hormonal contraception) or herbal remedies in the 14 days before IMP administration (See Section 11.4). Exceptions may apply on a case by case basis if considered not to interfere with the objectives of the study as agreed by the PI and sponsor's medical monitor
17. Use of any non-selective monoamine oxidase (MAO) inhibitors within 2 weeks of screening
18. History or presence of glaucoma
19. History or presence of suspicious undiagnosed skin lesions or a history of melanoma
20. Any history of psychoses or seizure
21. Known hypersensitivity to Sinemet® or domperidone or any of the excipients
22. Any history or presence of Prolactin-releasing pituitary tumour (prolactinoma)
23. Any medical history of GI haemorrhage, mechanical obstruction or perforation
24. Any history of moderate or severe hepatic impairment
25. Subjects with clinically significant liver function tests
26. Subjects with QTc >450 ms at screening
27. Subjects with significant electrolyte disturbances
28. Subjects with any underlying cardiac disease
29. Subjects who have received QT-prolonging drugs or potent cytochrome P450 (CYP) 3A4 inhibitors within 4 weeks of screening
30. ND0612H arm only: Subjects who have sinus problems
31. ND0612H arm only: Subjects who have regular heartburn and/or indigestion
32. ND0612H arm only: Subjects who have had abdominal (bowel) surgery
33. ND0612H arm only: Any clinically significant findings observed during naso-jejunal tube placement as determined by the endoscopist
34. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Cmax (maximal plasma concentration) of CD for different doses of CD | 6 days
  Pre-infusion and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 17, 20, 22, 24, 25, 26, 27, 28, 29, 30, 31, and 32 hours after commencing the ND0612 infusion on Days 1, 3 and 5.
AUC (area under the curve) of CD for different doses of CD | 6 days
  Pre-infusion and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 17, 20, 22, 24, 25, 26, 27, 28, 29, 30, 31, and 32 hours after commencing the ND0612 infusion on Days 1, 3 and 5.
Cmax (maximal plasma concentration) of LD and CD for ND0612 vs. LCIG | 4 days
  Pre-infusion and at 1, 2, 3, 4, 6, 9, 12, 14, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after commencing the LCIG infusion on Days 1 and 3.
AUC (area under the curve) of LD and CD for ND0612. LCIG | 4 days
  Pre-infusion and at 1, 2, 3, 4, 6, 9, 12, 14, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after commencing the LCIG infusion on Days 1 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Philip evans, MBChB, MRCS, Principal Investigator — Quotient Clinical LTD
Locations (1):
- Quotient Clinical LTD, Ruddington, Nottingham, United Kingdom